CLINICAL TRIAL: NCT03205657
Title: MAC and autoHSCT, Targeted Immunotherapy and RIC alloHSCT in Children, Adolescents, and Young Adults (CAYA) With Poor-risk Refractory/Relapsed Mature B-NHL: A Retrospective Chart Review
Brief Title: Auto/Allo Tandem Transplant for Relapsed B-NHL
Status: Completed | Type: Observational
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: L 11,813
Record Dates: First submitted 2017-05-11; First posted 2017-07-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: auto transplant followed by allo transplant — patients who got MAC conditioning with auto SCT followed by RIC followed by alloSCT for mature B-NHL

SUMMARY:
The investigators plan to perform a retrospective review of patients with poor risk relapsed/refractory B-NHL having received HSCT and targeted immunotherapy at the Maria Fareri Children's Hospital between January 1, 2012 and June 1, 2015. The investigators will review the clinical records and collect the data with de-identified medical information from our HSCT clinical research database.

DETAILED DESCRIPTION:
The investigators will obtain the following information from the patient's medical records: clinical factors including age at presentation, gender, clinical presentation, laboratory and pathology data, lymphoma diagnosis, clinical staging criteria, anti-cancer therapy as well as supportive care medicines, complications of therapy (adverse events graded from CTCAE v4.0), and hematopoietic stem cell transplantation therapy (chemotherapy, donor source, cell dose), course (engraftment, GVHD, chimerism), and follow-up (disease status).

ELIGIBILITY:
Inclusion Criteria:

* This analysis will include all children, adolescents, and young adults less than 29 years old with a histologically confirmed diagnosis of B-NHL treated at the Maria Fareri Children's Hospital

Exclusion Criteria:

* None

Ages: 0 Years to 29 Years | Sex: All
Age Groups: Child, Adult
Study Population: B-NHL patients who received MAC/AutoSCT and a RIC/AlloSCT
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to study treatment (safety) | 3 years
  Adverse events (according to CTCAE 4.0) will be reviewed for all as well as outcome data retrospectively to determine if the treatment was equal or better than standard of care for relapse/refractory B-NHL in terms of the number of adverse events reported. Data reviewed will include laboratory values, radiology exams and disease evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardenswartz A, Mehta B, El-Mallawany NK, van de Ven C, Hochberg J, Flower A, Morris E, Harrison L, Chu Y, Basso J, Gerard P, Islam H, Ayello J, Baxter-Lowe LA, Cairo MS. Safety and efficacy of combinatorial therapy utilizing myeloablative conditioning and autologous stem cell transplantation, targeted immunotherapy, and reduced intensity conditioning and allogeneic stem cell transplantation in children, adolescents, and young adults with relapsed/refractory mature B-cell non-Hodgkin lymphoma. Leuk Lymphoma. 2023 Jan;64(1):234-237. doi: 10.1080/10428194.2022.2133542. Epub 2022 Oct 19. No abstract available. PMID 36260003